CLINICAL TRIAL: NCT00235547
Title: Immediate Versus Delayed Initiation of Transdermal Hormonal Contraception After Therapeutic Abortion: A Randomized Trial
Brief Title: Trial of Immediate Versus Delayed Initiation of Transdermal Hormonal Contraception After Therapeutic Abortion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H11779-2703-01
Record Dates: First submitted 2005-10-06; First posted 2005-10-10 (Estimated); Results first posted 2019-06-10 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Abortion
Keywords: abortion; randomized; contraception; pregnancy; compliance; continuation; contraceptive patch; transdermal hormonal contraception
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- contraception-Immediate start (Active Comparator): contraception after abortion and before leaving the clinic, observed by clinic staff
  Interventions: Behavioral: timing of initiation of transdermal patch after an abortion
- Contraception-Delayed start (Active Comparator): instructed to begin contraception the first Sunday after leaving the clinic
  Interventions: Behavioral: timing of initiation of transdermal patch after an abortion

INTERVENTIONS:
Behavioral: timing of initiation of transdermal patch after an abortion — the initiation of the patch after abortion is dictated by the study as opposed to offering several options (i.e. first Sunday of period). For this arm it is to place the patch in the clinic with clinic staff before leaving the clinic

SUMMARY:
This is a randomized, controlled trial investigating whether immediate versus standard, "Sunday Start", initiation of transdermal hormonal contraception (the patch) in post-abortion subjects can improve compliance and the continuation of contraception. Immediate initiation of the patch has been studied in women seeking contraception when they are not immediately post-abortion, and this "Quick Start" method has been shown to improve the continuation of the patch into a second month. The primary hypothesis of this study is that immediate initiation of the patch in post-abortal women will improve the continuation of contraception over delayed initiation on the first Sunday after an abortion.

DETAILED DESCRIPTION:
The United States has a higher rate of unintended pregnancy than Canada or any other developed nation in Europe. Hormonal contraception is the most common method of contraception used in this country. Perfect use can lead to failure rates as low as 0.1% per year. Actual failure rates are much higher, often due to non-compliance with contraception use. Several recent studies have examined the "Quick Start", or initiation of hormonal contraception (OCPs and patch) in front of the provider while still at the clinic, regardless of time in the cycle. These studies have shown that women who placed the first patch in the clinic were more likely to continue the patch into the second month. Women who are seen in clinics for a therapeutic abortion (TAB) are often at extremely high risk for another unintended/unwanted pregnancy. If compliance in patch use could be improved in this group of women, unintended/unwanted pregnancy rates could be reduced. One concern about the "Quick Start" technique is that women may have already ovulated or conceived when the patch is initiated mid-cycle. In the post-abortal setting, this is not a concern. Applying the "Quick Start" technique to post-abortion patients and having women place the first patch while still in the clinic after their abortion may improve compliance and continuation of patch use.

This is a prospective, randomized, controlled trial in post-abortal women, and will last approximately 24 months. All of the study subjects will receive a month's worth of the patch and a one-year prescription after their TAB. The women in the immediate start arm will then place their first patch in the clinic, observed by clinic staff, before leaving. The controls will be instructed to place the first patch on the first Sunday following their abortion. All subjects will receive the same medication with the only difference being the timing of initiation of the patch. Measurements of continuation will be determined by telephone interviews administered at two and six months after the subjects' abortion.

ELIGIBILITY:
Inclusion Criteria:

* Any woman aged 13-45 who presents to the Women's Options Clinic and desires to use the patch for post-abortion contraception.

Exclusion Criteria:

* Gestational age above 23 weeks and 1 day.
* Any absolute contraindication for patch use (smoking > 20 cigarettes a day over age 35, history of venous thromboembolic event or pulmonary embolism, history of or current ischemic heart disease, history of stroke, vascular disease, complicated valvular heart disease [pulmonary hypertension, atrial fibrillation, history of subacute bacterial endocarditis], severe hypertension with blood pressure >160/100, migraines with focal neurologic symptoms, current breast cancer, active viral hepatitis, severe cirrhosis, or benign or malignant liver tumors).
* Patients who speak languages other than English or Spanish.
* Patients who do not have a phone or who have a phone where any contact might compromise the confidentiality of their abortions.

Ages: 13 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 298 (Actual)
Dates: Start 2005-08; Primary Completion 2006-05 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jody E Steinauer, MD, MAS, Principal Investigator — University of California, San Francisco; Sarah W Prager, MD, Study Director — University of California, San Francisco
Locations (1):
- Women's Options Clinic at San Francisco General Hospital, San Francisco, California, United States

REFERENCES:
- [Derived] Steinauer JE, Sokoloff A, Roberts EM, Drey EA, Dehlendorf CE, Prager SW. Immediate versus delayed initiation of the contraceptive patch after abortion: a randomized trial. Contraception. 2014 Jan;89(1):42-7. doi: 10.1016/j.contraception.2013.03.002. Epub 2013 Mar 13. PMID 24176251

RESULTS

PARTICIPANT FLOW:
Period: 2 Month Follow-up Survey
Arm/Group | Contraception-Immediate Start | Contraception-Delayed Start
Started | 154 | 144
Completed | 108 | 104
Not Completed | 46 | 40
Period: 6 Month Follow-up Survey
Arm/Group | Contraception-Immediate Start | Contraception-Delayed Start
Started | 154 | 144
Completed | 83 | 76
Not Completed | 71 | 68

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Contraception-Immediate Start | Contraception-Delayed Start | Total
Number analyzed (Participants) | 154 | 144 | 298
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.9 (5.3) | 22.5 (5.2) | 22.2 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 154 | 144 | 298
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Latina | 53 | 47 | 100
  Race/Ethnicity: African-American | 46 | 45 | 91
  Race/Ethnicity: White | 25 | 26 | 51
  Race/Ethnicity: Asian/PI | 24 | 24 | 48
  Race/Ethnicity: Multiracial/Other | 6 | 2 | 8
Insurance [Count of Participants; unit: Participants]
  Medi-Cal/Emergency Medi-CAl | 124 | 118 | 242
  Private or HMO | 11 | 5 | 16
  Self-pay | 19 | 21 | 40
BMI [Mean (Standard Deviation); unit: BMI] | 25.0 (4.5) | 24.9 (4.0) | 24.9 (4.3)
Prior patch use [Count of Participants; unit: Participants] | 53 | 54 | 107

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Use Patch After Abortion, by Study Arm
Description: we will also describe what participants were using two months post-abortion
Time Frame: six months after enrollment/abortion
Population: randomized subjects who completed the six month survey
Measure: Count of Participants; unit: Participants
Arm/Group | Contraception-Immediate Start | Contraception-Delayed Start
Number analyzed (Participants) | 83 | 76
Participants | 36 | 42

2. Secondary Outcome: Number of Participants Who Were Using Effective Method at 6 Months Post-enrollment
Description: An effective method is defined as a hormonal method or intra-uterine device
Time Frame: six months post enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Contraception-Immediate Start | Contraception-Delayed Start
Number analyzed (Participants) | 83 | 76
Participants | 46 | 49

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Contraception-Immediate Start | Contraception-Delayed Start
Serious Adverse Events (participants affected / at risk) | 0/154 | 0/144
Other Adverse Events (participants affected / at risk) | 0/154 | 0/144

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No